CLINICAL TRIAL: NCT00179699
Title: Phase I Open-Label, Dose Escalation Study To Determine The Maximum Tolerated Dose And To Evaluate The Safety Profile Of Lenalidomide (Revlimid®, CC-5013) With Pemetrexed In Subjects With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NSCL-002
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2005-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: cc-5013; Non Small Cell Lung Cancer; revlimid; celgene; cc5013
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Lenalidomide; Pemetrexed

INTERVENTIONS:
Drug: CC-5013
Drug: pemetrexed

SUMMARY:
Study will deteremine the MTD and evaluate the safety profile of oral lenalidomide on days 1-14 when combined with pemetrexed on day 1 of a 21 days cycle. Subjects will continue on study until documention of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and voluntarily sign an informed consent document.
2. Age >or= 18 years at the time of signing informed consent form.
3. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
4. Histological or cytologic documentation of advanced NSCLC.
5. Radiographic or clinical evidence of measurable advanced NSCLC. Subjects must have measurable disease at least 2 cm in diameter.
6. Subjects must have been treated and progressed following chemotherapy.
7. ECOG performance status of 0 or 1 (Appendix I: ECOG Performance Status Scale).
8. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000 cells/mm3 (100 x 109/L)
   3. Serum creatinine >1.5 mg/dL (133 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >or = 1.5 mg/dL (26 mmol/L)
2. Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent.
3. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the breast) unless the subject has been free of disease for > 1 year.
4. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
5. More than one prior chemotherapy for advanced NSCLC.
6. Concurrent use of any other anti-cancer agents.
7. Any prior use of lenalidomide.
8. Pregnant or lactating females.
9. Prior > or = to grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
10. Prior > or = to grade 3 allergic reaction/hypersensitivity to thalidomide.
11. Use of any standard/experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy.
12. Known Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09; Study Completion 2006-11

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and evaluate the safety profile of oral lenalidomide on days 1-14 and pemetrexed on day 1 every 21 days, as combination therapy to subjects with advanced Non-Small Cell Lung Cancer

SECONDARY OUTCOMES:
To explore the anit-tumor activity of the combination of lenalidomide and pemetrexed when given to subjects with advanced NSCLC

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - MD Anderson - Orlando, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - North Shore Hem/Onc Associates, East Setauket, New York